CLINICAL TRIAL: NCT05908890
Title: A Study to Determine the Efficacy of a Denture Adhesive Formulation to Seal Out Food Particles From Under the Mandibular Partial Denture
Brief Title: A Study to Determine the Efficacy of a Denture Adhesive to Seal Out Food Particles From Under the Mandibular Partial Denture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 2018129
Record Dates: First submitted 2023-06-05; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Partial Denture

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Denture Adhesive (Experimental)
  Interventions: Device: Experimental Denture Adhesive
- Marketed Denture Adhesive (Active Comparator)
  Interventions: Device: Fixodent True Feel Denture Adhesive

INTERVENTIONS:
Device: Experimental Denture Adhesive — Adhesive will be applied to the partial denture(s) by a dental professional separate from the examiner and subject.
  Arms: Experimental Denture Adhesive
Device: Fixodent True Feel Denture Adhesive — Adhesive will be applied to the partial denture(s) by a dental professional separate from the examiner and subject.
  Arms: Marketed Denture Adhesive

SUMMARY:
The objective of this study is to evaluate the effectiveness of two denture adhesives at keeping food particles (seeds) from becoming trapped underneath partial denture(s).

ELIGIBILITY:
Inclusion Criteria:

* give written informed consent prior to their participation;
* be 18 years of age or older;
* have a Kennedy Class I or class II partial mandibular denture with a minimum of three consecutive teeth on the prosthesis;
* have a history of food particles getting under their partial, mandibular denture;
* agree not to use any denture adhesive on the day of their study visits, prior to the visit;
* agree to not participate in any other oral/dental product studies during the study;
* be willing to use or not use denture adhesive as instructed during the treatment periods;
* be willing to eat a poppy seed muffin;
* be in good general health as determined by the Investigator/designee based on a review of the medical history/update; and
* have a minimum of 4 total poppy seeds on their mandibular denture base and gingiva after eating the muffin.

Exclusion Criteria:

* present with any disease or conditions that could be expected to interfere with examination procedures or the subject's safe completion of the study;
* self-report that they are allergic to denture adhesives or to the test food (gluten intolerance to muffin or intolerance to poppy seeds); or
* have appliances with intracorneal attachments, crowns with precision attachments or implant overdentures:
* have any condition or medication which, in the opinion of the investigator, is currently causing xerostomia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2019-10-03 (Actual); Study Completion 2019-10-03 (Actual)

PRIMARY OUTCOMES:
Poppy Seed Count Before Treatment Application | Immediately following consumption of the muffin before treatment application
  Subjects ate 1/2 top of a poppy seed muffin. After eating the muffin, subjects were instructed to remove their partial mandibular denture and a dental professional counted the number of poppy seeds remaining on the subject's partial denture base and gingiva.
Poppy Seed Count After Treatment Application | Immediately following consumption of the muffin after treatment application
  Subjects ate 1/2 top of a poppy seed muffin. After eating the muffin, subjects were instructed to remove their partial mandibular denture and a dental professional counted the number of poppy seeds remaining on the subject's partial denture base and gingiva.

CONTACTS AND LOCATIONS:
Locations (1):
- Salus Research, Inc, Fort Wayne, Indiana, United States